CLINICAL TRIAL: NCT02613962
Title: A Prospective, Multicentric Clinical Proof-of-concept Study to Stratify Targeted Therapies Adapted to Molecular Profiling of Relapsed or Refractory Pediatric Tumors
Brief Title: Proof -of -Concept Study To Stratify Targeted Therapies Adapted To Molecular Profiling
Acronym: MAPPYACTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Innovative Therapies For Children with Cancer Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2015-A00464-45; 2015/2244 (Other: CSET number)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Relapsed or Refractory Pediatric Tumor
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- relapsed or refractory pediatric tumor (Experimental): This is a prospective, international, multicentric clinical proof-of-concept study to stratify targeted therapies adapted to molecular profiling of relapsed or refractory pediatric tumors. The molecular screening will be done on a newly biopsied or resected tumor sample obtained at the time of relapse/progression, using high-throughput technologies, primarily WES and RNA Sequencing, and bioinformatics analysis.
  Interventions: Procedure: biopsy or surgical resection of tumor and blood sampling

INTERVENTIONS:
Procedure: biopsy or surgical resection of tumor and blood sampling

SUMMARY:
In the light of the development of high-throughput technologies enabling a biology-based reclassification of tumors and the increasing number of available specifically targeting anticancer agents the era of "precision medicine" has begun. Several clinical precision medicine trials with the aim of stratifying treatment according to molecular profiles (for example in France: 'MOlecular Screening for CAncer Treatment Optimization' MOSCATO-01, SHIVA, PROFILER, Safir01, Safir02) are ongoing in adults and have shown the feasibility of this approach. MOSCATO-01 is the first trial worldwide including pediatric patients, performing an on-purpose intervention and molecular profiling in recurrent tumors. Together with more than 500 adult patients, between December 2012 to August 2014, the tumors of 35 children and adolescents have been profiled, confirming that this approach is feasible in pediatric patients albeit with accelerated time stringencies. Importantly, the results of the first children and adolescents profiled showed that 2/3 of patients had 'actionable' alterations using hot spot mutations sequencing and CGH array (Geoerger B et al, ASCO 2014).

The project 'MAPPYACTS' will use both Whole Exome Sequencing (WES) and RNA Sequencing of tumor tissue to increase the number of targetable genomic alterations. Furthermore to improve understanding of the overall molecular profile and possible response to treatment, methylation array, miRNA expression profiles, and study of immunomodulators will be performed on tumor samples subsequently. CLIP2 (INCa-labeled early phase clinical trials centers) - SiRIC (INCa- labeled comprehensive cancer centers) molecular profiling and bioinformatics platforms will contribute with their expertise in molecular profiling projects and characterization of pediatric cancers. Data interpretation of molecular genetic alterations detected by WES and RNA Seq and treatment recommendation will be done within a multidisciplinary therapeutic molecular biology tumor board.

'MAPPYACTS' will produce one of the largest cohorts of molecularly characterized relapsed tumors reported to date, and thanks to increased access to clinical trials since the European pediatric legislation, the investigators expect that 20-30% of patients can be stratified into a targeted trial based on the detected profile.

It is the investigators' intention that this initiative paves the way to enrich ongoing clinical targeted agent trials, to increase the numbers of stratified clinical trials, to an earlier access to targeted agents, and will play a crucial role in the relevant development of these new agents in pediatric malignancies.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent signed by the patient, or parents or legal representative and assent of the minor child to perform biopsy/surgical resection/aspiral/sample and molecular analysis of the tumor and blood sample
* Patient with confirmed solid tumor or leukemia which is recurrent or refractory to standard treatment and who is eligible for an early phase clinical trial
* In case of solid tumor, lesion must be accessible for biopsy or surgical resection or cytological puncture
* Age: Patients aged ≥ 6 months at time of inclusion and aged ≤ 18 years at the time of initial diagnosis
* Performance status and life expectancy that allows treatment in an experimental trial: Karnofsky performance status ≥ 70% for patients > 12 years of age, Lansky play scale ≥ 70% for patients ≤ 12 years of age
* Adequate organ function:

Adequate hematopoietic function for patients with solid tumor (Leukemia patients are excluded from hematological criteria) : Neutrophils >1.0 x 109/l, Platelets >100 x 109/l, Heamoglobin >80 g/l (transfusion allowed) In case of bone marrow involvment: Neutrophils >/= 0.75 x 109/l (unsupported) , Platelet count >/= 0.75 x 109/l (unsupported) Adequate hepatic function: ALAT/ASAT <2.5 x ULN, Bilirubin ≤1.5 x ULN (in case of tumor involvement of the liver ALAT/ASAT <5 x ULN) Adequate renal function: Serum creatinemia <1.5 x ULN for age. In case serum creatinine >1.5 ULN according to age, creatinine clearance has to be >70mL/mL/1.73 m2 or glomerular filtration rate measurement >70% of the expected value

- Patients affiliated to a Social Security Regimen or beneficiary of the same as per local regulatory requirements

Exclusion criteria:

* Life expectancy ≤ 3 months
* Symptomatic CNS metastases
* In case of leukemia, are excluded patients with isolated meningitis relapses.
* Coagulation disorder that prevents the accomplishment of a biopsy or surgery
* Uncontrolled infections not responsive to antibiotics, antiviral medicines, or antifungal medicines
* Presence of ≥ CTCAE grade 2 toxicity (except alopecia, ototoxicity, lymphopenia which are not excluded if grade 3 or less) due to prior cancer therapy
* Malignant disease other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 3 years prior to study entry
* Any concurrent illness or laboratory abnormality that in opinion of investigator may interfere with the interpretation of study results, may suppose a risk for the realization of biopsy/surgery, and in the judgment of the investigator would make the patient inappropriate for the study
* Evidence of active viral Hepatitis B or C or known diagnosis of human immunodeficiency virus infection

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 700 (Estimated)
Dates: Start 2016-01-13 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with recurrent or refractory pediatric solid tumor or leukemia that could be attributed to treatment with matched targeted agents | assessed four years after beginning of study
  The percentage of patients with recurrent or refractory pediatric solid tumor or leukemia that could be attributed to treatment with matched targeted agents according to the molecular profile in their individual tumor will be estimated

CONTACTS AND LOCATIONS:
Locations (5):
- Gustave Roussy, Villejuif, Val De Marne, France
- Our Lady's Children's Hospital, Dublin, Crumlin, Ireland
- Schneider Children's Medical Center, Petah Tikva, Israel
- Fondazione IRCCS Istituto, Milan, Italy
- Hospital Universitari Vall D'Hebron, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Chaix J, Schleiermacher G, Corradini N, Andre N, Thebaud E, Gambart M, Defachelles AS, Entz-Werle N, Chastagner P, De Carli E, Ducassou S, Landman-Parker J, Adam-de-Beaumais T, Larive A, Michiels S, Vassal G, Valteau-Couanet D, Geoerger B, Berlanga P. Clinical trial inclusion in patients with relapsed/refractory neuroblastoma following the European Precision Cancer Medicine trial MAPPYACTS. Eur J Cancer. 2024 Apr;201:113923. doi: 10.1016/j.ejca.2024.113923. Epub 2024 Feb 15. PMID 38377775
- [Derived] Marques Da Costa ME, Zaidi S, Scoazec JY, Droit R, Lim WC, Marchais A, Salmon J, Cherkaoui S, Morscher RJ, Laurent A, Malinge S, Mercher T, Tabone-Eglinger S, Goddard I, Pflumio F, Calvo J, Redini F, Entz-Werle N, Soriano A, Villanueva A, Cairo S, Chastagner P, Moro M, Owens C, Casanova M, Hladun-Alvaro R, Berlanga P, Daudigeos-Dubus E, Dessen P, Zitvogel L, Lacroix L, Pierron G, Delattre O, Schleiermacher G, Surdez D, Geoerger B. A biobank of pediatric patient-derived-xenograft models in cancer precision medicine trial MAPPYACTS for relapsed and refractory tumors. Commun Biol. 2023 Sep 18;6(1):949. doi: 10.1038/s42003-023-05320-0. PMID 37723198
- [Derived] Berlanga P, Pierron G, Lacroix L, Chicard M, Adam de Beaumais T, Marchais A, Harttrampf AC, Iddir Y, Larive A, Soriano Fernandez A, Hezam I, Chevassus C, Bernard V, Cotteret S, Scoazec JY, Gauthier A, Abbou S, Corradini N, Andre N, Aerts I, Thebaud E, Casanova M, Owens C, Hladun-Alvaro R, Michiels S, Delattre O, Vassal G, Schleiermacher G, Geoerger B. The European MAPPYACTS Trial: Precision Medicine Program in Pediatric and Adolescent Patients with Recurrent Malignancies. Cancer Discov. 2022 May 2;12(5):1266-1281. doi: 10.1158/2159-8290.CD-21-1136. PMID 35292802
- [Derived] Morscher RJ, Brard C, Berlanga P, Marshall LV, Andre N, Rubino J, Aerts I, De Carli E, Corradini N, Nebchi S, Paoletti X, Mortimer P, Lacroix L, Pierron G, Schleiermacher G, Vassal G, Geoerger B. First-in-child phase I/II study of the dual mTORC1/2 inhibitor vistusertib (AZD2014) as monotherapy and in combination with topotecan-temozolomide in children with advanced malignancies: arms E and F of the AcSe-ESMART trial. Eur J Cancer. 2021 Nov;157:268-277. doi: 10.1016/j.ejca.2021.08.010. Epub 2021 Sep 17. PMID 34543871
- [Derived] Peneder P, Stutz AM, Surdez D, Krumbholz M, Semper S, Chicard M, Sheffield NC, Pierron G, Lapouble E, Totzl M, Erguner B, Barreca D, Rendeiro AF, Agaimy A, Boztug H, Engstler G, Dworzak M, Bernkopf M, Taschner-Mandl S, Ambros IM, Myklebost O, Marec-Berard P, Burchill SA, Brennan B, Strauss SJ, Whelan J, Schleiermacher G, Schaefer C, Dirksen U, Hutter C, Boye K, Ambros PF, Delattre O, Metzler M, Bock C, Tomazou EM. Multimodal analysis of cell-free DNA whole-genome sequencing for pediatric cancers with low mutational burden. Nat Commun. 2021 May 28;12(1):3230. doi: 10.1038/s41467-021-23445-w. PMID 34050156